CLINICAL TRIAL: NCT02283723
Title: Health Teams Advancing Patient Experience: Strengthening Quality (TAPESTRY): A Randomized Controlled Trial Using the Health TAPESTRY Approach to Care for Older Adults
Brief Title: A Randomized Controlled Trial Using the Health TAPESTRY Approach to Care for Older Adults
Acronym: HealthTAPESTRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Health Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 14-726
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Aging
Keywords: older adults, goal attainment, optimal aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Group 1 (Experimental): This patient group will begin receiving the Health TAPESTRY intervention from time zero.
  Interventions: Other: Health TAPESTRY Intervention
- Patient Group 2 (Active Comparator): Using a step-wedge approach, this patient group will receive the intervention after a six month waiting period where they will be used as a comparable group. In the first six months, they will receive usual care.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Health TAPESTRY Intervention — The patient will receive in-home visits from trained volunteers to assess overall health and wellness and discover any health goals patient might have. This information will be electronically communicated back to interprofessional healthcare team and used to create informed care plan, link to relevant community services and allow the patient to age optimally.
  Arms: Patient Group 1
Other: Usual care — While waiting for the Health TAPESTRY intervention, the control group will receive usual care from their healthcare providers.
  Arms: Patient Group 2

SUMMARY:
Health TAPESTRY is a delayed intervention pragmatic randomized control trial promoting interprofessional team collaboration, facilitating connection to the community through system navigation and trained community volunteers, enhancing communication and improving care through the use of technology to better understand and assist older adult patients in achieving their health goals and to enable them to have optimal aging.

DETAILED DESCRIPTION:
The overarching aim of the integrated multicomponent Health TAPESTRY approach is to promote optimal aging. Optimal aging within the Health TAPESTRY program means supporting people to move through life with good health in the best possible way: Being Alive Well. Health TAPESTRY is a health and social care approach that centres on meeting a person's health goals with the support of technology, trained community volunteers, an interprofessional team, system navigation, and better links between primary care and community organizations. The Health TAPESTRY intervention takes a complex, multilevel approach to integration, from both system level and individual level perspectives. The Health TAPESTRY program will provide processes and tools to activate and support individuals to access and use the broad range of available primary health care, social and community services to achieve their personal health goals and strategies to better integrate care at the system level. More specifically Health TAPESTRY will promote optimal aging:

* through intentional, proactive conversations about a person's life, health and care goals within the primary healthcare setting;
* through improved connections between inter-professional primary care teams, community service providers and informal caregivers;
* by training volunteers to serve as a link between the primary care team and a person in their home;
* by using technology from the home to link directly with the primary health care team which includes
* the tablet-based Health TAPESTRY app for volunteers to use;
* the Personal Health Record (PHR) and
* innovative resources (i.e. Optimal Aging Portal).

It is anticipated that together these will enable transformation of how primary healthcare and interprofessional teams provide care to older adults in a manner that provides value for resources used and meets needs and goals of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Any community-dwelling patient of McMaster Family Health Team over the age of 70

Exclusion Criteria:

* Patient is palliative or receiving end-of-life care
* Patient is deceased
* Has explicitly stated that they do not want to be part of a research project
* Patient resides in long-term care
* Patient has indicated that they do not want to receive a home visit from trained community volunteers.
* Patient or family member does not speak English
* Patient will be out of the country for more than 50% of trial duration

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 316 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Progress attaining health goals | 12 months
  The participant will identify up to 5 areas of health that will serve as the basis for Goal Attainment Scale(GAS) measurement and will assign subjective weights using a scale of 1 to 9 (higher scores indicating greater importance). An indicator for each goal is selected and used to indicate progress in meeting the goal. The expected outcomes for each problem area will be identified. These outcomes will be standardized and as descriptive, objective and observable as possible. The indicators will be applied to the intervention group and control group in the same manner. Participants will be followed up at the end of 6 months by an independent and blinded assessor for the purpose of study comparison to evaluate the patient's level of goal attainment for each priority problem area that has a goal attainment scale constructed for it although participants in the intervention group may have follow occur more frequently as the information about goals is transmitted to the health care team

SECONDARY OUTCOMES:
Quality of life measures (2 tools) | 12 months
  1)The EuroQol-5 Demensop-5 Level (EQ-5D-5L) is comprised of six questions investigating patients' present health status. The last question requires patients to rate one's own current health status on a scale from 0-100, 0 being worst and 100 being the best; and 2)Veterans Rand-12 (VR-12) It's a 9 item survey that focuses mainly on physical and emotional health. The survey was developed at RAND Corporation with the support of US Department of Veterans Affairs. Both of these tools are under consideration by the Canadian Institute of Health Research (CIHR) led community based primary healthcare indicators group and the proposed TAPESTRY study offers the opportunity to compare the two tools.
Self-efficacy Scale | 12 months
  The scale measures the ability and confidence of patient to self-manage their own health. The scale comprises of 6 items and each item is responded on a 10-point Likert scale with 0 indicates not at all confident and 10 denotes totally confident.
Optimal aging | 12 months
  Single question, "In terms of your own healthy aging, would you say it is excellent, very good, good, fair, or poor?" Ratings become a 5-point scale ranging from 1 to 5. A similar question has been used in the Canadian Longitudinal Study on Aging.
Duke Social Support Index | 12 months
  This validated scale is comprised of 11 questions. The first seven questions measure satisfaction with social support and the latter five questions assess social networking. Satisfaction score range from 6-18 whereas networking scores ranges from 4-12. The scale facilitates understanding patients' relationships with friends/family and whoever supports them. Those individuals who score less than 10 on the satisfaction scale are considered at risk.
Comprehensiveness | 12 months
  Perceived clinic comprehensives regarding patient healthcare needs will be assessed via CIHR common indicator (comprehensiveness domain). Participants respond to 4 questions using a 4-point scale ("not at all" to "definitely"), with an additional option of "I haven't needed such support.
Patient Empowerment | 12 months
  The extent to which participants feel in control with regard to healthcare is measure via CIHR common indicator (patient empowerment domain). Participants respond to 5 questions using a 4-point scale ("not at all" to "definitely").
Patient Centredness | 12 months
  The extent to which participants feel their healthcare team addresses what matters to them will be assessed via CIHR common indicator (Patient-Centredness domain). Participants respond to 6 questions using a 4-point scale ("not at all" to "completely").
Access | 12 months
  Patient access to services will be assessed via CIHR common indicators project: Access subdomain.
Satisfaction with Care | 12 months
  This is a one item scale that about satisfaction with primary care received. Participants are asked to rate their level of satisfaction from 1 ("not at all satisfied") to 10 ("completely satisfied").
Hospitalizations for Ambulatory Care Sensitive Conditions (ACSC) for Chronic Disease | 12 months
  An indirect measure of access to primary care is seen for example, in increased for diagnoses that can be effectively managed outside hospital (ambulatory care sensitive conditions; ACSCs). ACSCs such as chronic obstructive pulmonary diseases, asthma, diabetes, hypertension, angina and others), have rates of 387 per 100,000 for those aged 75 to 84 years compared to 2240 per 100,000 for those 85 years or older. Hospitalizations for Adverse Events will also be calculated.
Caregiver Strain Index | 12 months
  For those participant who answer "yes" to being a caregiver, the 4-item Zarit screen will be administered in addition to a description of the context of their caregiving will be given. For this screen, participants answer 4 questions using a 5-point scale from "never" to "always".
Cost-effectiveness | 12 months
  Program costs: Will be measured using micro costing techniques where a healthcare cost and Resource utilization form has been pilot tested to record resources used during the implementation of the TAPESTRY program. This resource use information will be combined with unit prices for each resource and summed across all resources to estimate the total cost of the program. Maintaining and updating infrastructure costs will be included. Healthcare resource use and cost: Will be obtained from the patient questionnaire that will assess cost and resources involved in providing healthcare for older adults.

OTHER OUTCOMES:
Patients' Satisfaction with Volunteers | 12 months
  Patients will be asked to rate their level of satisfaction with volunteer visits.
Team Functioning | 12 months
  An adapted version of the Organizational Readiness for Change Assessment (ORCA) will be used to measure team functioning. This questionnaire includes 18 questions to assess evidence, context, and facilitation and to give a general sense of healthcare professionals' perceptions of the clinic's organizational readiness for change as it relates to the uptake of TAPESTRY
Volunteers' Self-efficacy | 12 months
  Volunteers will be asked to rate their confidence in performing 3 tasks related to a volunteer visit for each visit they complete.

CONTACTS AND LOCATIONS:
Overall Officials: David Price, MD, Study Chair — McMaster University
Locations (2):
- Canada (2):
  - McMaster Family Practice, Hamilton, Ontario
  - Stonechurch Family Health Centre, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaber J, Oliver D, Valaitis R, Cleghorn L, Lamarche L, Avilla E, Parascandalo F, Price D, Dolovich L. Experiences of integrating community volunteers as extensions of the primary care team to help support older adults at home: a qualitative study. BMC Fam Pract. 2020 May 16;21(1):92. doi: 10.1186/s12875-020-01165-2. PMID 32416718
- [Derived] Valaitis R, Cleghorn L, Dolovich L, Agarwal G, Gaber J, Mangin D, Oliver D, Parascandalo F, Ploeg J, Risdon C. Examining Interprofessional teams structures and processes in the implementation of a primary care intervention (Health TAPESTRY) for older adults using normalization process theory. BMC Fam Pract. 2020 Apr 15;21(1):63. doi: 10.1186/s12875-020-01131-y. PMID 32295524
- [Derived] Dolovich L, Oliver D, Lamarche L, Thabane L, Valaitis R, Agarwal G, Carr T, Foster G, Griffith L, Javadi D, Kastner M, Mangin D, Papaioannou A, Ploeg J, Raina P, Richardson J, Risdon C, Santaguida P, Straus S, Price D. Combining volunteers and primary care teamwork to support health goals and needs of older adults: a pragmatic randomized controlled trial. CMAJ. 2019 May 6;191(18):E491-E500. doi: 10.1503/cmaj.181173. PMID 31061074
- [Derived] Dolovich L, Oliver D, Lamarche L, Agarwal G, Carr T, Chan D, Cleghorn L, Griffith L, Javadi D, Kastner M, Longaphy J, Mangin D, Papaioannou A, Ploeg J, Raina P, Richardson J, Risdon C, Santaguida PL, Straus S, Thabane L, Valaitis R, Price D. A protocol for a pragmatic randomized controlled trial using the Health Teams Advancing Patient Experience: Strengthening Quality (Health TAPESTRY) platform approach to promote person-focused primary healthcare for older adults. Implement Sci. 2016 Apr 5;11:49. doi: 10.1186/s13012-016-0407-5. PMID 27044360